CLINICAL TRIAL: NCT07355972
Title: A Clinical Study Exploring the Safety, Efficacy and Cellular Metabolic Dynamics of CT1195E Car-t Cell Injection in Refractory / Progressive Systemic Sclerosis (SSC)
Brief Title: Safety, Efficacy and Cellular Metabolic Dynamics of CT1195E in Patients With Refractory / Progressive SSC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1195E-CG11010
Record Dates: First submitted 2025-11-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: SSc-Systemic Sclerosis
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT1195E CAR-T cells Injection (Experimental): CT1195E cells infusion
  Interventions: Other: CAR-T Therapy

INTERVENTIONS:
Other: CAR-T Therapy — CT1195E cells infusion

SUMMARY:
This study is a single arm, open label, exploratory dose escalation clinical study to evaluate the safety, efficacy, and cellular metabolic dynamics of ct1195e cells in patients with SSc.

The study was divided into dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily sign the informed consent form (ICF): I fully understand and know this study and sign the informed consent form. I am willing to follow and be able to complete all research procedures;
* when signing ICF, the age is between 18 and 60 years old (including 18 and 60 years old), regardless of gender;
* no systemic active infection (such as infectious pneumonia and tuberculosis) within 2 weeks before screening;
* women with fertility (defined as all women who are physically able to conceive) must agree to use efficient contraceptive methods from at least 28 days before the start of gonorrhea to 1 year after ct1195e infusion, and it is absolutely prohibited to donate eggs within 1 year after receiving study treatment infusion during the study period. Men whose partners are fertile must agree to use effective barrier contraception from the beginning of gonorrhea to 1 year after ct1195e infusion, and should not donate semen or sperm during the entire study period;
* women with fertility must be tested negative for serum β human chorionic gonadotropin (β -hcg) at the time of screening and within 48 hours before gonorrhea treatment.
* meet the 2013 eular/acr classification criteria for systemic sclerosis, and meet the diffuse manifestations, and the disease duration is ≤ 7 years (the onset time of the disease duration is defined as the time of the initial diagnosis of SSC);
* complicated with interstitial pneumonia, that is, the interstitial changes of ground glass exudation suggested by chest HRCT;
* meet the following definitions of refractory or progressive disease:

  1. Definition of refractory: the conventional treatment for more than 6 months is still ineffective, or the disease relapses after remission. Definition of conventional treatment: use of glucocorticoids (more than 1 mg/kg/d) or cyclophosphamide, as well as one or more of the following immunomodulatory drugs: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents, including yamerol, rituximab, belizumab, etanercept, etc;
  2. According to the definition of progressiveness, 2 of the following three items can be met in the past 1 year (within the past 1 year):

     1. Aggravation of symptoms;
     2. FVC estimated value decreases by 5%, or DLCO estimated value decreases by 10%;
     3. Pulmonary imaging aggravated;
* important organ functions:

  1. Renal function: defined as creatinine clearance (Cockcroft Gault) ≥ 50 ml/min calculated without hydration assistance;
  2. Bone marrow function: defined as neutrophil (ANC) ≥ 1.0 × 109/l, hemoglobin (HB) ≥ 90 g/l. Blood transfusion and growth factors shall not be used to meet the above requirements within 7 days before the eligibility screening;
  3. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × upper limit of normal (ULN), total bilirubin ≤ 2 × upper limit of normal (ULN)
  4. Coagulation function: INR ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN;
  5. Cardiac function: good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥ 40%.

Exclusion Criteria:

* FVC ≤ 30% predicted value or DLCO (corrected by hemoglobin) ≤ 30% predicted value;
* study participants with severe kidney disease or signs of renal crisis;
* there is active tuberculosis risk during screening: there are signs or symptoms of active tuberculosis judged by the investigator (such as fever, cough, night sweat and weight loss); Records of chest imaging (e.g., chest X-ray, chest CT scan) performed at screening or any time within 6 months before screening showed active tuberculosis.
* have previously received car-t cell or other gene modified T cell therapy, or have a history of major organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell / bone marrow transplantation;
* have used drugs targeting B cells (such as rituximab) within 3 months before screening;
* allergic or intolerant to Qinglin drugs and tocilizumab, or life-threatening allergic reaction, hypersensitivity reaction or intolerance to ct1195e preparation or its excipients (including dimethyl sulfoxide (DMSO), or previous history of other serious allergies such as allergic shock;
* prednisone (≥ 10 mg / day) (or equivalent drug) is used for hormones within 2 weeks before ct1195e infusion, and physiological replacement, local and inhalation hormones are allowed;
* received immunosuppressants affecting T cells (mycophenolate mofetil, methotrexate, cyclosporine, azathioprine, leflunomide, tacrolimus) within 2 weeks before infusion of ct1195e;
* received JAK inhibitors (tofacitinib, baricitinib tablets, lucotinib, etc.) within 2 weeks before ct1195e infusion;
* have been vaccinated with live attenuated vaccine, inactivated vaccine or RNA vaccine within 1 month before screening;
* suffering from malignant tumor within 2 years before signing ICF. Except for the following cases: non melanoma skin cancer after radical treatment, local prostate cancer, cervical carcinoma in situ confirmed by biopsy or squamous intraepithelial lesions detected by cervical smear, and breast carcinoma in situ that has been completely removed;
* major surgery has been performed within 4 weeks before signing the informed consent, or major surgery is planned to be required during the study, which the investigator believes will bring unacceptable risks to the study participants;
* HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (HCV antibody and HCV-RNA positive) were present at the time of screening;
* those with CNS diseases before screening include but are not limited to: cerebrovascular accident, encephalitis, epilepsy, convulsion / convulsion, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, CNS vasculitis, cognitive dysfunction, cerebral organic syndrome or psychosis;
* have a history of any of the following cardiovascular diseases within 1 month before screening: Grade III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia or other heart disease with significant clinical significance as defined by the New York Heart Association (NYHA);
* participate in other clinical studies within 3 months before screening or still within five half lives after the last medication.
* there is currently any uncontrollable active infection, including but not limited to active tuberculosis;
* if there is a history of suicidal thoughts or evidence within 6 months before signing the ICF, or any suicidal behavior within 12 months before signing the ICF, the investigator believes that there is a significant risk of suicide;
* pregnant or lactating women;
* the investigator judged that the study participants had poor compliance, were unable or unwilling to comply with the requirements of the study protocol, or were not suitable to participate in the clinical study for other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerable dose (MTD) and / or dose range of CT1195E were evaluated | After medication to day 28
  CT1195E MTD and/or dose range
severity of dose limiting toxicity (DLT) | Within 28 days after infusion
severity of adverse events (AES) | Within 180 days after infusion
Incidence of adverse events (AES) | Within 180 days after infusion
Incidence of dose limiting toxicity (DLT) | Within 28 days after infusion

SECONDARY OUTCOMES:
Changes of systemic sclerosis comprehensive response index score (acr-criss) from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The score range of the comprehensive response index for systemic sclerosis (acr-criss) is usually 0 to 100, where 0 represents the lowest disease activity and burden, and 100 represents the highest. The higher the score, the higher the disease activity, severity of skin involvement or overall disease burden of systemic sclerosis.
Changes from baseline in scleroderma clinical trials Association injury index (sctc-di) | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The minimum value of scleroderma clinical trials Association injury index (sctc-di) is 0 and the maximum value is 42. The higher the score, the more serious the organ damage, that is, the worse the result.
Changes from baseline in modified Rodnan skin scale (MRSS) | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The minimum value of the modified Rodnan skin scale (MRSS) is 0 points, and the maximum value is 57 points. The higher the score, the more severe the degree of skin sclerosis, that is, the worse the result. MRSS quantifies the skin involvement of systemic sclerosis by evaluating the skin hardness of 19 parts of the body. 0 points represent normal skin and 3 points represent severe thickening. The higher the total score, the more extensive and severe skin fibrosis, which is associated with disease activity and poor prognosis.
Changes in lung function (FVC) from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The normal value of FVC in healthy adults usually ranges from 3 to 5 liters, and the specific value varies according to age, sex, height, race and other factors. Higher FVC values usually indicate better lung function, because higher FVC means greater lung volume and stronger respiratory muscle strength.
Changes from baseline in left ventricular ejection fraction (LVEF) by cardiac function tests | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Changes of joint disease activity score (DAS-28) (if joint involvement) from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The minimum value of joint disease activity score (DAS-28) is 0 and the maximum value is 10. The higher the score, the higher the disease activity, that is, the worse the result, because the score is used to measure the activity of joint inflammation, and the increase of the score reflects the enhanced disease activity.
Changes of inflammation related indicators (CRP or ESR) from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
SSC specific antibodies (changes in anti-Scl-70 antibody levels from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Changes of anti RNA polymerase III antibody [rp155, rp11] levels from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Immune related autoantibodies (antinuclear antibody ANA) levels and changes from baseline | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Proportion of patients without other SSC therapies after medication | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Vascular lesions were assessed by nailfold capillary microscopy after medication | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Skin elasticity was assessed by skin ultrasound after medication | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Changes of chest HRCT in study participants after medication evaluation | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
Change from baseline in the post medication Health Assessment Questionnaire Disability Index (HAQ-DI) | 2 months and other time points after medication (the 1st, 3st, 6th, 9th and 12th months)
  The score range of the Health Assessment Questionnaire Disability Index (HAQ-DI) is usually 0 to 3, where 0 represents no disability or functional integrity, and 3 represents severe disability or inability to complete activities. The higher the score, the worse the patient's functional status, because HAQ-DI quantifies the degree of disability by evaluating the ability of daily activities, for example, the increased score in items such as dressing and walking reflects the increased difficulty.
The level of CT1195e transgene copy number in blood | Within 1 year after CAR-T cell infusion
Changes of B cell functional subsets (initial B cells, memory B cells, plasma cells) after ct1195E infusion | Within 1 year after CAR-T cell infusion
Duration of ct1195e transgene copy number in blood | Within 1 year after CAR-T cell infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospita, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No